CLINICAL TRIAL: NCT02394769
Title: ASPIRED: ASPirin Intervention for the REDuction of Colorectal Cancer Risk
Brief Title: ASPirin Intervention for the REDuction of Colorectal Cancer Risk
Acronym: ASPIRED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew T. Chan, MD, MPH, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-496; R01CA137178 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (For Aspirin) (Placebo Comparator): The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy (start of randomization). Participants will be expected to take one capsule orally at the blinded dose, once daily, until the final visit. Duration not to exceed 12 weeks.
  Interventions: Drug: Placebo for Aspirin
- Low Dose Aspirin (Active Comparator): The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy (start of randomization). Participants will be expected to take one capsule orally at the blinded dose (81 mg/d), once daily, until the final visit. Duration not to exceed 12 weeks.
  Interventions: Drug: Aspirin
- Standard Dose Aspirin (Active Comparator): The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy (start of randomization). Participants will be expected to take one capsule orally at the blinded dose (325mg/d), once daily, until the final visit. Duration not to exceed 12 weeks.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin
  Other Names: 2-Acetylsalicylic Acid; ASA
  Arms: Low Dose Aspirin; Standard Dose Aspirin
Drug: Placebo for Aspirin
  Arms: Placebo (For Aspirin)

SUMMARY:
This research study is investigating the use of aspirin as a potential chemopreventive agent to reduce risk of colorectal cancer

DETAILED DESCRIPTION:
This research study, is investigating the use of aspirin as a potential chemopreventive agent to reduce risk of colorectal cancer. Within the gastroenterology practice of Massachusetts General Hospital (MGH), we will conduct a prospective, double-blind, placebo-controlled, randomized clinical trial to measure the effects of daily low-dose (81 mg/day) and standard-dose (325 mg/day) aspirin on urine, plasma, stool, and tissue biomarkers associated with colorectal cancer.

Aspirin is part of the non-steroidal anti-inflammatory drug (NSAID) family, which are drugs routinely used for their pain-killing (analgesic), fever-reducing (antipyretic), or anti-inflammatory properties. Most NSAIDs are available as over-the-counter formulations. Substantial evidence has conclusively demonstrated that aspirin reduces the risk of colorectal neoplasia, yet there remains uncertainty surrounding its mode of action. Aspirin has already been established to reduce the risk of cardiovascular disease. Prospective studies as well as randomized clinical trials demonstrate that aspirin reduces the risk of precancerous polyps and colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Underwent screening or surveillance colonoscopy at MGH within the last 9 months with removal of at least one adenoma.
* Age 18-80 years.
* This study will only include adult participants because colorectal carcinogenesis in children is more likely to be related to a cancer predisposition syndrome with distinct biological mechanisms compared with sporadic colorectal cancer in adults. Patients over age 80 will not be enrolled since the benefits and risks of a daily aspirin regimen over the age of 80 have not yet been well-characterized.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Not currently taking aspirin (any dose) within the last 6 months.
* The effects of aspirin on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Use of any non-aspirin non-steroidal anti-inflammatory drug (NSAID) at any dose at least three times a week during the two months prior to randomization.
* Diagnosis of inflammatory bowel disease, liver or kidney disease, bleeding diathesis
* Any prior diagnosis of gastrointestinal cancer (including esophageal, small intestine, colon, pancreatic), or any diagnosis of other cancers (with the exception of non- melanoma skin) in which there has been any active treatment within the last three years
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aspirin.
* Known diagnosis of Familial Adenomatous Polyposis (FAP) or Hereditary Non-Polyposis Colorectal Cancer (HNPCC, Lynch Syndrome).
* Any adenoma that was not completely removed during previous colonoscopy.
* History of aspirin intolerance, bleeding diathesis, peptic ulcer or gastrointestinal bleed, endoscopic complications, or contraindication to colonoscopy.
* Inability or unwillingness to abstain from non-protocol use of aspirin or NSAIDs or to provide blood, urine, or stool samples or colon biopsies during the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding.
* Pregnant women are excluded from this study because aspirin is an FDA Category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with aspirin, breastfeeding should be discontinued if the mother is treated with aspirin.
* Participant must be able to swallow pills.
* Participant is taking any anticoagulant agent (e.g. warfarin) or antiplatelet agent (e.g. clopidogrel).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2029-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Chan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Drew DA, Chin SM, Gilpin KK, Parziale M, Pond E, Schuck MM, Stewart K, Flagg M, Rawlings CA, Backman V, Carolan PJ, Chung DC, Colizzo FP 3rd, Freedman M, Gala M, Garber JJ, Huttenhower C, Kedrin D, Khalili H, Kwon DS, Markowitz SD, Milne GL, Nishioka NS, Richter JM, Roy HK, Staller K, Wang M, Chan AT. ASPirin Intervention for the REDuction of colorectal cancer risk (ASPIRED): a study protocol for a randomized controlled trial. Trials. 2017 Feb 1;18(1):50. doi: 10.1186/s13063-016-1744-z. PMID 28143522
- [Background] Drew DA, Schuck MM, Magicheva-Gupta MV, Stewart KO, Gilpin KK, Miller P, Parziale MP, Pond EN, Takacsi-Nagy O, Zerjav DC, Chin SM, Mackinnon Krems J, Meixell D, Joshi AD, Ma W, Colizzo FP, Carolan PJ, Nishioka NS, Staller K, Richter JM, Khalili H, Gala MK, Garber JJ, Chung DC, Yarze JC, Zukerberg L, Petrucci G, Rocca B, Patrono C, Milne GL, Wang M, Chan AT. Effect of Low-dose and Standard-dose Aspirin on PGE2 Biosynthesis Among Individuals with Colorectal Adenomas: A Randomized Clinical Trial. Cancer Prev Res (Phila). 2020 Oct;13(10):877-888. doi: 10.1158/1940-6207.CAPR-20-0216. Epub 2020 Jul 27. PMID 32718943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who meet the inclusion criteria will be identified through investigators during their routine clinical practice, supplemented by a periodic query of the MGH endoscopy and pathology databases. Potentially eligible participants are approached by letter from their treating physician. Two weeks after receiving the letter, study staff will contact eligible parties and screen for eligibility via phone interview. Enrollment began in July 2015 and ended in February 2019.
Groups:
- Placebo (For Aspirin): The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy (start of randomization). Participants will be expected to take one capsule orally at the blinded dose, once daily, until the final visit. Duration not to exceed 12 weeks.
  Placebo for Aspirin
- Low Dose Aspirin: The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy (start of randomization). Participants will be expected to take one capsule orally at the blinded dose (81 mg/d), once daily, until the final visit. Duration not to exceed 12 weeks.
  Aspirin
- Standard Dose Aspirin: The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy (start of randomization). Participants will be expected to take one capsule orally at the blinded dose (325mg/d), once daily, until the final visit. Duration not to exceed 12 weeks.
  Aspirin
Period: Overall Study
Arm/Group | Placebo (For Aspirin) | Low Dose Aspirin | Standard Dose Aspirin
Started | 60 | 60 | 60
Completed | 58 | 57 | 54
Not Completed | 2 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (For Aspirin) | Low Dose Aspirin | Standard Dose Aspirin | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.2) | 56.1 (8.7) | 57.5 (8.3) | 56.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 28 | 85
  Male | 32 | 31 | 32 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 58 | 58 | 59 | 175
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 3 | 10
  White | 55 | 52 | 53 | 160
  More than one race | 0 | 4 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1
Marital status [Count of Participants; unit: Participants]
  Married | 40 | 39 | 37 | 116
  Never married | 6 | 12 | 11 | 29
  Separated | 2 | 0 | 1 | 3
  Divorced | 8 | 7 | 7 | 22
  Widowed | 4 | 2 | 4 | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.8 (5.0) | 28.4 (4.9) | 27.5 (5.7) | 27.6 (5.2)
Body Mass Index, categories [Count of Participants; unit: Participants]
  Normal, <18.5-24.9 | 21 | 16 | 21 | 58
  Overweight, 25.0-29.9 | 26 | 26 | 23 | 75
  Obese ≥30.0 | 13 | 18 | 16 | 47
Smoking status [Count of Participants; unit: Participants]
  Never | 38 | 36 | 32 | 106
  Former | 18 | 20 | 19 | 57
  Current | 4 | 3 | 8 | 15
  Missing | 0 | 1 | 1 | 2
Alcohol consumption [Count of Participants; unit: Participants]
  Never | 7 | 11 | 11 | 29
  Rarely | 14 | 16 | 18 | 48
  1-5 times/week | 29 | 24 | 23 | 76
  Daily | 10 | 8 | 6 | 24
  More than daily | 0 | 1 | 2 | 3
Personal cancer history, yes [Count of Participants; unit: Participants] | 10 | 6 | 4 | 20
Family history of colorectal cancer, yes [Count of Participants; unit: Participants] | 13 | 10 | 12 | 35
Type II diabetes, yes [Count of Participants; unit: Participants] | 2 | 3 | 2 | 7
Menopause status [Number; unit: participants] — Population: Menopausal status of female participants, only
  participants
    Premenopausal: number analyzed (Participants) | 28 | 29 | 28 | 85
    Premenopausal | 3 | 9 | 5 | 17
    Perimenopausal: number analyzed (Participants) | 28 | 29 | 28 | 85
    Perimenopausal | 4 | 1 | 2 | 7
    Postmenopausal: number analyzed (Participants) | 28 | 29 | 28 | 85
    Postmenopausal | 20 | 17 | 18 | 55
    Missing: number analyzed (Participants) | 28 | 29 | 28 | 85
    Missing | 1 | 2 | 3 | 6
History of 81 mg aspirin use [Count of Participants; unit: Participants]
  Never | 55 | 50 | 53 | 158
  Intermittently (<2x/week) | 2 | 5 | 5 | 12
  Regularly (>2x/week) | 2 | 2 | 2 | 6
  Missing | 1 | 3 | 0 | 4
History of 325 mg aspirin use [Count of Participants; unit: Participants]
  Never | 40 | 42 | 42 | 124
  Intermittently (<2x/week) | 17 | 15 | 17 | 49
  Regularly (>2x/week) | 1 | 1 | 1 | 3
  Missing | 2 | 2 | 0 | 4
History of non-steroidal anti-inflammatory drug use [Count of Participants; unit: Participants]
  Never | 18 | 13 | 19 | 50
  Intermittently (<2x/week) | 31 | 36 | 32 | 99
  Regularly (>2x/week) | 10 | 9 | 8 | 27
  Missing | 1 | 2 | 1 | 4
Proton pump inhibitor use [Count of Participants; unit: Participants]
  Current and regular | 5 | 6 | 8 | 19
  No, never regularly | 48 | 49 | 48 | 145
  Missing | 7 | 5 | 4 | 16
H2-blocker use [Count of Participants; unit: Participants]
  Current and regular | 2 | 5 | 2 | 9
  No, never regularly | 56 | 54 | 57 | 167
  Missing | 2 | 1 | 1 | 4
Antacid use [Count of Participants; unit: Participants]
  Current and regular | 5 | 3 | 3 | 11
  No, never regularly | 54 | 57 | 57 | 168
  Missing | 1 | 0 | 0 | 1
Statin use [Count of Participants; unit: Participants]
  Current and regular | 14 | 11 | 16 | 41
  No, never regularly | 44 | 48 | 43 | 135
  Missing | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Prostaglandin Metabolites (PGE-M)
Description: Measured using liquid chromatography/mass spectrometry
Time Frame: 8-12 weeks
Measure: Mean (Standard Deviation); unit: ng/mg cr
Arm/Group | Placebo (For Aspirin) | Low Dose Aspirin | Standard Dose Aspirin
Number analyzed (Participants) | 58 | 57 | 54
ng/mg cr
  Baseline urinary PGE-M | 15.5 (12.6) | 17.7 (17.1) | 14.3 (13.7)
  Post-intervention urinary PGE-M | 16.4 (15.8) | 13.1 (13.4) | 9.4 (7.9)
  Change in urinary PGE-M | 0.8 (11.8) | -4.6 (17.7) | -4.9 (11.2)

2. Secondary Outcome: Plasma Macrophage Inhibitory Cytokine-1 (MIC-1), an Inflammatory Biomarker
Description: Measured using an ELISA for MIC-1
Time Frame: 8-12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Chromatin Binding
Description: Measured using ChIP-Seq of DNA extracted from colonic epithelium
Time Frame: 8-12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Expression of Wnt-associated Signaling Genes (CTNNB1, AXIN2 and MYC)
Description: Measured using RNA-seq of colonic epithelium
Time Frame: 8-12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Spectral Biomarkers of Colorectal Cancer
Description: Measured using Partial Wave Spectroscopy on rectal cytology brushing samples
Time Frame: 8-12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo (For Aspirin) | Low Dose Aspirin | Standard Dose Aspirin
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 14/60 | 17/60 | 17/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (For Aspirin) (N=60) | Low Dose Aspirin (N=60) | Standard Dose Aspirin (N=60)
GI upset (i.e. heartburn/acid reflux/nausea/gas) (Gastrointestinal disorders) | 4 | 6 | 3
Unrelated infection/cold symptoms/sinus related (General disorders) | 6 | 5 | 4
Extended bleeding/bruising (Blood and lymphatic system disorders) | 0 | 0 | 2
Bleeding hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Seasonal allergies (General disorders) | 1 | 2 | 3
Fever (General disorders) | 1 | 0 | 2
Headaches (Nervous system disorders) | 0 | 1 | 0
Other, unrelated (General disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02394769/Prot_SAP_000.pdf